CLINICAL TRIAL: NCT02218281
Title: Developing a Smartphone App With Mindfulness Training for Teen Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Lori Pbert, Professor of Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R34DA037886 (NIH)
Record Dates: First submitted 2014-07-29; First posted 2014-08-18 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- C2Q-Teen app (Experimental): Smoking cessation treatment delivered through a smartphone app via mindfulness training.
  Interventions: Behavioral: C2Q-Teen app
- NCI's QuitSTART app (Active Comparator): Smoking cessation treatment delivered through a smartphone app by NCI, without mindfulness training.
  Interventions: Behavioral: NCI's QuitSTART app
- Written smoking cessation materials only (Active Comparator): Receipt of written smoking cessation materials.
  Interventions: Behavioral: Written smoking cessation materials only

INTERVENTIONS:
Behavioral: C2Q-Teen app — Commit to Quit (C2Q)-Teen app provides smoking cessation assistance incorporating mindfulness training.
  Arms: C2Q-Teen app
Behavioral: NCI's QuitSTART app — NCI's smoking cessation app
  Arms: NCI's QuitSTART app
Behavioral: Written smoking cessation materials only — Receipt of written smoking cessation materials
  Arms: Written smoking cessation materials only

SUMMARY:
The recent Surgeon General's Report calls for effective and readily available treatment approaches to help adolescent smokers interested in quitting. Schools are an ideal venue for connecting adolescent smokers with smoking cessation assistance. This study will adapt the Craving to Quit (C2Q) smartphone app, which integrates mindfulness training into a smoking cessation program, for teen smokers (C2Q-Teen). We will test how well this novel app helps teens stop smoking compared to another teen smoking cessation app that does not include mindfulness training, and to written cessation information alone. If effective, the C2Q-Teen would be relatively easy to disseminate widely and have tremendous public health significance

DETAILED DESCRIPTION:
The new Surgeon General's Report (SGR), Preventing Tobacco Use Among Youth and Young Adults, highlights the addictive nature of nicotine and emphasizes the need for effective and accessible cessation treatment for the more than 3.6 million youth who smoke. This proposal is in response to PA-13-078, Behavioral and Integrative Treatment Development Program (R34), which supports the development and testing of behavioral interventions targeting substance abuse, including studies focused on Intervention generation and refinement (Stage IA), and pilot or feasibility (Stage IB), and research designed to "increase implementability of interventions with creative use of technology". We have developed Craving to Quit (C2Q), a smartphone intervention for smoking cessation for adults that integrates mindfulness training (MT) into a smoking cessation curriculum. While MT has been shown to be efficacious for smoking cessation in adults, it has not been tested in adolescents. In addition, dissemination of MT is challenging due to the need for experienced MT therapists, high time demand, difficulties in scheduling sessions, and high costs of in-person treatment delivery. Mobile, smartphone technologies provide a promising medium for overcoming these barriers to dissemination. We propose to adapt and refine our existing Craving to Quit (C2Q) app for use by adolescent smokers (Stage IA), and to conduct feasibility and pilot testing (Stage IB) in preparation for an R01 application to definitively test efficacy and probe psychological mechanisms of change resulting from MT. In the pilot test, six public high schools will be randomly assigned to one of three conditions, two schools per condition: (1) C2Q-Teen app (smoking cessation delivered through a smartphone app via MT), (2) NCI's QuitSTART app designed for teen smokers (NCI-QS) (smoking cessation delivered through a smartphone app without MT), or (3) written smoking cessation materials only (MO). One hundred forty four adolescent smokers interested in quitting will be recruited (24/school, 48/condition). School nurses will introduce the three interventions in the school setting. Our first primary aim is to adapt the C2Q app for use by adolescent smokers (C2Q-Teen). Our second primary aim is to evaluate the feasibility and acceptability of the interventions to ensure adequacy of each intervention for a larger RCT designed specifically to compare efficacy rates. Secondary aims are to assess relative efficacy of the three interventions and independent contributions of smartphone intervention delivery and mindfulness in increasing cotinine-validated 7-day point prevalence abstinence at 3- and 6-month follow-up in order to adequately power a larger trial, and to determine the relationship between C2Q-Teen usage and abstinence. If eventually found to be effective, C2Q-Teen offers an innovative and potentially powerful intervention for supporting teens in their efforts to quit that would be relatively easy to disseminate widely and have tremendous public health significance, addressing the SGR's call for readily available treatment for adolescent smokers wanting to quit

ELIGIBILITY:
Inclusion Criteria:

* enrolled in grade 9-12
* smoked at least 5 cigarettes on average per day for the past 7 days
* interested in quitting smoking in the next three weeks
* have a smartphone on iPhone or Android platforms
* English-speaking

Exclusion Criteria:

* unable or unwilling to provide informed assent
* diagnosis of a serious psychiatric illness during the past 5 years
* developmental delay that would prevent study participation

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of study recruitment into the three interventions | Baseline
  We will assess the ability to recruit 144 adolescents into the trial at baseline.
Feasibility of retention of participants at 3-month follow-up | 3-month follow-up
  We will assess the ability to retain 80% of the 144 adolescents recruited at 3-month follow-up.
Feasibility of retention of participants at 6-month follow-up | 6-month follow-up
  We will assess the ability to retain 80% of the 144 adolescents recruited at 6-month follow-up.
Acceptability of the three interventions | 3-month follow-up
  Assess the percentage of participants in each condition that indicate high utilization and acceptability ratings (at least 80% hypothesized)

SECONDARY OUTCOMES:
Cotinine-validated 7-day point prevalence abstinence | 3- and 6-months follow-up
  Self-reported 7-day point abstinence confirmed by cotinine. Saliva samples will be collected from all participants prior to survey completion at each follow-up assessment. Samples will be analyzed for cotinine for all subjects reporting abstinence for the past 7 days. We will use cotinine-validated abstinence (cut-off of 11.4 ng/ml) and a cotinine-imputed abstinence when cotinine is missing.
C2Q-Teen program usage as a predictor of smoking abstinence | 3- and 6-month follow-up
  It is hypothesized that C2Q-Teen program usage, defined as self-report of the number of C2Q-Teen modules completed and informal mindfulness practice, will predict smoking abstinence at 3-month follow-up and at 6-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Pbert, PhD, Principal Investigator — University of Massachusetts, Worcester; Judson Brewer, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- [Derived] Pbert L, Druker S, Crawford S, Frisard C, Trivedi M, Osganian SK, Brewer J. Feasibility of a Smartphone App with Mindfulness Training for Adolescent Smoking Cessation: Craving to Quit (C2Q)-Teen. Mindfulness (N Y). 2020 Mar;11(3):720-733. doi: 10.1007/s12671-019-01273-w. Epub 2019 Dec 20. PMID 33343761